CLINICAL TRIAL: NCT04288778
Title: A Prospective, Multi-centric, Open-label, Single-arm, Phase 4 Study to Evaluate the Safety and Efficacy of Canagliflozin + Metformin Hydrochloride IR Fixed-dose Combination as an Adjunct to Diet and Exercise to Improve Glycemic Control in Indian Adult Patients With Type 2 Diabetes Mellitus When Treatment With Both Canagliflozin and Metformin is Appropriate
Brief Title: A Study to Assess Safety of Canagliflozin and Metformin Hydrochloride Combination Given as a Supplement to Diet and Exercise to Improve Blood Sugar Level in Indian Adult Participants With Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108749; 28431754DIA4032 (Other: Johnson & Johnson Private Limited)
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Results first posted 2023-08-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Canagliflozin; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Canagliflozin + Metformin Hydrochloride Immediate Release (IR) (Experimental): Participants will receive canagliflozin + metformin hydrochloride IR fixed-dose combination, 50 milligram (mg) + 500 mg or 50 mg + 1000 mg, will be provided as tablets for oral administration.
  Interventions: Drug: Canagliflozin + Metformin hydrochloride (Fixed Dose Combination)

INTERVENTIONS:
Drug: Canagliflozin + Metformin hydrochloride (Fixed Dose Combination) — Participants will receive canagliflozin + metformin hydrochloride IR fixed-dose combination, 50 milligram (mg) + 500 mg or 50 mg + 1000 mg, will be provided as tablets for oral administration. The study Treatment duration will be of 24 weeks.
  Other Names: JNJ-28431754

SUMMARY:
The purpose of this study is to assess safety of canagliflozin + metformin hydrochloride immediate Release (IR) fixed-dose combination.

ELIGIBILITY:
Inclusion Criteria:

* Participant willing to adhere to diet and exercise regimen as recommended by the investigator
* Type 2 diabetes mellitus (T2DM) with inadequate glycemic control on diet and exercise, who in investigator's opinion are eligible to receive study drug as per prescribing information along with standard care for management of T2DM
* Women must be postmenopausal, defined as greater than (>) 45 years of age with amenorrhea for at least 18 months, or > 45 years of age with amenorrhea for at least 6 months and less than (<) 18 months and a serum follicle stimulating hormone (FSH) level > 40 International Units Per Liter (IU/L), or surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal occlusion), or otherwise be incapable of pregnancy, or sexually active and practicing a highly effective method of birth control, including hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, tubal ligation, intrauterine device, double-barrier method (example, condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), or male partner sterilization, and consistent with local regulations regarding use of birth control methods for participant participating in clinical studies, for the duration of their participation in the study, or not sexually active
* Women of childbearing potential, regardless of age must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and negative UPT at baseline (predose, Day 1)
* Treatment naive participants or participants on stable antihyperglycemic agent (AHA) therapy (for at least 12 weeks before screening) and have a screening visit Glycosylated Haemoglobin (HbA1c) of greater than or equal to (>=) 7.0 percent (%) and less than or equal to (<=) 10.0 %

Exclusion Criteria:

* History of liver or renal insufficiency (estimated creatinine clearance below 45 milliliter per minute [mL/min]); significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Known allergies, hypersensitivity, or intolerance to Canagliflozin, Metformin or Canagliflozin + metformin hydrochloride immediate release (IR) Fixed Dose combination (FDC) or its excipients
* Use of any other sodium glucose cotransporter 2 (SGLT2) inhibitor within 12 weeks before the screening visit
* If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days after last dose of study medication; or intending to donate ova during such time period
* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Private Limited Clinical Trial, Study Director — Johnson & Johnson Private Limited
Locations (10):
- India (10):
  - Lifecare Hospital and Research Centre, Bengaluru
  - Post Graduate Institute of Medical Education And Research PGIMER, Chandigarh
  - Kovai Diabetes Specialty Centre & Hospital, Coimbatore
  - Excelcare Hospitals (A unit of Asclepius Hospitals and Health Care Pvt. Ltd.), Guwahati
  - Thumbay Hospital New life / Endocrinology, Hyderabad
  - Fortis Hospital, Mohali
  - Jehangir Clinical Development Center Pvt Ltd, Pune
  - Chellaram Diabetes Institute, Pune
  - Nirmal Hospital Pvt. Ltd., Surat
  - Jothydev's Diabetes Research Centre, Trivandrum

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] LaRoche JK, Lanier J, Alvarenga R, Collins M, Costelloe T, Chiau A, Whetherly H, De Soete W, Faludi J, Rens K. Climate footprint of industry-sponsored in-human clinical trials: life cycle assessments of clinical trials spanning multiple phases and disease areas. BMJ Open. 2025 Feb 19;15(2):e085364. doi: 10.1136/bmjopen-2024-085364. PMID 39971605

RESULTS

PARTICIPANT FLOW:
Groups:
- Canagliflozin + Metformin Hydrochloride FDC: Participants received either (canagliflozin 50 milligram [mg] + metformin hydrochloride 500 mg) or (canagliflozin 50 mg + metformin hydrochloride 1000 mg) immediate release (IR) fixed-dose combination (FDC) tablets twice daily (BD) up to Week 24.
Period: Overall Study
Arm/Group | Canagliflozin + Metformin Hydrochloride FDC
Started | 276
Treated | 274
Completed | 265
Not Completed | 11
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 5
Not completed — Non-Compliance With Study Drug | 1
Not completed — Other | 1
Not completed — Started but not treated | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had taken at least 1 dose of study treatment.
Arm/Group | Canagliflozin + Metformin Hydrochloride FDC
Number analyzed (Participants) | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 168
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indian | 274
Region of Enrollment [Count of Participants; unit: Participants]
  India | 274

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was any untoward medical occurrence that at any dose resulted in death, was life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product. TEAEs were defined as events that started on or after the study medication start date and time.
Time Frame: Baseline (Day 1) up to 24 weeks
Population: Safety analysis set included all participants who had taken at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Canagliflozin + Metformin Hydrochloride FDC
Number analyzed (Participants) | 274
Percentage of participants
  TEAEs | 41.6
  TESAEs | 1.1

2. Primary Outcome: Percentage of Participants With Unexpected Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An adverse event was considered unexpected if the nature or severity was not consistent with the applicable product reference safety information.
Time Frame: Baseline (Day 1) up to 24 weeks
Population: Safety analysis set included all participants who had taken at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Canagliflozin + Metformin Hydrochloride FDC
Number analyzed (Participants) | 274
Percentage of participants | 0

3. Secondary Outcome: Percent Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Weeks 12 and 24
Description: Percent change from baseline in HbA1c at Weeks 12 and 24 was reported.
Time Frame: Baseline, Weeks 12 and 24
Population: Efficacy analysis set included all participants who had taken at least 1 dose of study treatment and had both baseline and at least 1 post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) represents number of participants evaluable at the specified timepoints.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Canagliflozin + Metformin Hydrochloride FDC
Number analyzed (Participants) | 265
Percent change
  Percent change at Week 12: number analyzed (Participants) | 264
  Percent change at Week 12 | -0.918 (1.1348)
  Percent change at Week 24 | -0.926 (1.3054)

4. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs)
Description: ADRs were defined as the treatment related TEAEs. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. TEAEs were defined as events that started on or after the study medication start date and time.
Time Frame: Baseline (Day 1) up to 24 weeks
Population: Safety analysis set included all participants who had taken at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Canagliflozin + Metformin Hydrochloride FDC
Number analyzed (Participants) | 274
Percentage of participants | 10.6

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to end of study (28 weeks)
Description: Safety analysis set included all participants who had taken at least 1 dose of study treatment.
Arm/Group | Canagliflozin + Metformin Hydrochloride FDC
All-Cause Mortality (participants affected / at risk) | 0/274
Serious Adverse Events (participants affected / at risk) | 3/274
Other Adverse Events (participants affected / at risk) | 114/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin + Metformin Hydrochloride FDC (N=274)
COVID-19 (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1
Prostatomegaly (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin + Metformin Hydrochloride FDC (N=274)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Hydrocele (Congenital, familial and genetic disorders) | 1
Cataract (Eye disorders) | 1
Diabetic Retinal Oedema (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Hyperchlorhydria (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 5
Chest Pain (General disorders) | 1
Fatigue (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 13
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 5
Carbuncle (Infections and infestations) | 1
Dengue Fever (Infections and infestations) | 2
Dysentery (Infections and infestations) | 1
Fungal Infection (Infections and infestations) | 2
Fungal Skin Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Genital Infection (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 2
Orchitis (Infections and infestations) | 1
Tinea Cruris (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 7
Vaginal Infection (Infections and infestations) | 1
Vulvovaginitis (Infections and infestations) | 1
Limb Injury (Injury, poisoning and procedural complications) | 1
Albumin Urine Present (Investigations) | 4
Blood Creatinine Increased (Investigations) | 1
Blood Pressure Increased (Investigations) | 1
Blood Triglycerides Increased (Investigations) | 3
Urine Albumin/Creatinine Ratio Increased (Investigations) | 2
Weight Decreased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 13
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 9
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 4
Dizziness Exertional (Nervous system disorders) | 1
Head Discomfort (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 1
Albuminuria (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 3
Microalbuminuria (Renal and urinary disorders) | 3
Micturition Urgency (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 5
Adenomyosis (Reproductive system and breast disorders) | 1
Balanoposthitis (Reproductive system and breast disorders) | 4
Prostatomegaly (Reproductive system and breast disorders) | 1
Pruritus Genital (Reproductive system and breast disorders) | 1
Smegma Accumulation (Reproductive system and breast disorders) | 1
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Pruritus (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT04288778/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT04288778/SAP_001.pdf